CLINICAL TRIAL: NCT03526328
Title: Doublecortin Like Kinase-1 as a Marker and Indicator of Treatment Response for Intestinal Stem Cells in Barrett's Esophagus and Progression to Esophageal Adenocarcinoma
Brief Title: DCLK1 as a Marker/Indicator of Stem Cell Response in Barrett's Esophagus/Esophageal Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 1885
Record Dates: First submitted 2013-09-26; First posted 2018-05-16 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Barrett's Esophagus; Esophageal Adenocarcinoma
Keywords: DCLK1; Serum Biomarker; Barrett's Esophagus; Esophageal Adenocarcinoma; Tumor Stem Cell Marker
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DCLK1 post BE treatment: Effects of EMR and RFA on the expression of putative stem cell biomarkers and correlate them with serum/plasma protein expression and disease progression and/or recurrence (Barrett's esophagus/ esophageal adenocarcinoma)
  Interventions: Other: EMR and RFA effect on stem cell marker expression in BE/EAC

INTERVENTIONS:
Other: EMR and RFA effect on stem cell marker expression in BE/EAC — Observation of EMR and RFA on the expression of putative stem cell biomarkers and correlate them with serum/plasma protein expression and disease progression and/or recurrence (Barrett's esophagus/ esophageal adenocarcinoma)

SUMMARY:
The hypotheses are: 1) the intestinal stem cell marker, DCLK1, which is increased in both the epithelium and stroma in colon cancer is also increased in BE (Barrett's esophagus) with HGD (high grade dysplasia) and in EAC (esophageal adenocarcinoma), 2) this expression correlates with disease progression towards EAC and 3) eradication of cells expressing stem cell markers occurs after therapy of EMR (endoscopic mucosal resection) or RFA (radiofrequency ablation) to eradicate BE with HGD and intramucosal adenocarcinoma and esophagectomy for EAC. We will test our hypotheses with the following aims: 1) To characterize the cell specific expression patterns of intestinal stem cell biomarkers in BE patients and correlate them with serum expression and disease progression, 2) To examine prospectively the effects of EMR, RFA or esophagectomy on the expression of stem cell biomarkers and the progression to EAC.

DETAILED DESCRIPTION:
Barrett's esophagus (BE) is a metaplasia of normal squamous epithelium. BE can progressively develop more abnormal features like low-grade intraepithelial dysplasia (LGID), high-grade intraepithelial dysplasia (HGID) before ultimately developing esophageal adenocarcinoma (EAC), with a low 5-year survival rate of 20 % or less. Recent evidence for the existence of cancer stem cells (CSCs) has advanced our understanding of cancer and has opened doors to new therapeutic strategies in cancer treatment. The fundamental goals of this project are to determine the effectiveness of endoscopic mucosal resection (EMR) and radiofrequency ablation (RFA) on eradication of putative intestinal stem cell markers that are overexpressed in BE with HGID and EAC. A better understanding of the cellular mechanisms that regulate the progression from normal squamous mucosa to EAC has enormous implications in the diagnosis and treatment of esophageal cancer. The presence of a CSC in esophageal cancer has been reported in both dysplastic BE/ EAC as well as in mouse models of the disease. The central hypotheses of the current proposal are: elimination of cells expressing stem cell markers occurs after ablative therapies (EMR/RFA) to eradicate BE with HGID/ EAC, and monitoring of stem cell marker expression during follow-up will correlate with disease recurrence or appropriate clinical response. Recently, we have reported that DCLK1, although minimally expressed in normal distal esophageal squamous mucosa, is markedly expressed in BE epithelium and EAC. We will test our central hypotheses with the following specific aims: 1. To prospectively characterize the cell specific expression patterns of putative intestinal stem cell biomarkers in BE patients and correlate them with serum/plasma protein expression and disease progression, 2. to examine prospectively the effects of EMR/RFA on the expression of putative stem cell biomarkers and correlate them with serum/plasma protein expression and disease progression and/or recurrence, and 3. to examine prospectively the effects on EMR/ RFA on esophageal-related quality of life and dysphagia during the endoscopic intervention period as well as following completion. The studies proposed have the potential to offer new insights for both the early diagnosis and monitoring of therapeutic response of future therapies for EAC. Moreover, these studies may identify novel biomarkers that can aid in the confirmation of HGID and potentially predict disease onset, progression and/or recurrence. Finally, these studies have the potential to provide preliminary data that will serve as the rationale for large scale multicenter trials to compare the effectiveness of EMR and RFA in BE with respect to clinical outcome, molecular features and effect on putative tumor stem cells. The recent identification of DCLK1 as a marker that distinguishes between normal and tumor stem cells in a rodent model of intestinal tumorigenesis lends support for our rationale for examining DCLK1 as a potential mediator of the neoplastic response in BE.

ELIGIBILITY:
Inclusion Criteria:

* BE length of 12 cm or less
* presence of non-dysplastic BE on 2 sequential endoscopies or low-grade intraepithelial dysplasia (LGIN), high-grade intraepithelial dysplasia (HGIN) or EAC in BE segment on 2 endoscopies in the previous 6 months
* no signs of metastasis on endoscopic ultrasonography or computerized tomography scan.

Exclusion Criteria:

* pre-RFA EMR with cancer at the resection margin
* greater than T1sm1 invasion
* poor differentiation or worse
* angiolymphatic invasion
* esophageal stenosis preventing passage of an 11.3 mm endoscope
* persistent visible lesions after EMR before RFA and invasive cancer on biopsies after EMR pre-RFA.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for upper endoscopy to evaluate symptoms or risk factors such as GERD, dyspepsia, or dysphagia with a finding of BE or EAC; treatment with EMR or RFA for BE with HGD, focal intramucosal adenocarcinoma or esophagectomy for EAC.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-03; Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
cell-specific expression patterns of putative intestinal stem cell biomarkers in BE patients; correlation of markers with serum/plasma protein expression and disease progression. | 2 yrs
  Exploratory; analysis of expression of various markers for Barrett's esophagus and esophogeal adenocarcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Bolkhir, MD, Principal Investigator — University of Oklahoma
Locations (1):
- Gastroenterology, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Background] Vega KJ, May R, Sureban SM, Lightfoot SA, Qu D, Reed A, Weygant N, Ramanujam R, Souza R, Madhoun M, Whorton J, Anant S, Meltzer SJ, Houchen CW. Identification of the putative intestinal stem cell marker doublecortin and CaM kinase-like-1 in Barrett's esophagus and esophageal adenocarcinoma. J Gastroenterol Hepatol. 2012 Apr;27(4):773-80. doi: 10.1111/j.1440-1746.2011.06928.x. PMID 21916995